CLINICAL TRIAL: NCT01753856
Title: Anabolism Versus Antiresorption: A Quadruple Labeling Histomorphometry Study to Compare the Mechanism of Action of Teriparatide and Denosumab in Postmenopausal Women With Osteoporosis
Brief Title: Effects of Teriparatide or Denosumab on Bone in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14592; B3D-US-GHDV (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-18; First posted 2012-12-20 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Denosumab; Demeclocycline; Tetracycline; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): 20 micrograms (µg) teriparatide administered subcutaneously (SC) once every day for 6 months.
  Demeclocycline (DEM): Beginning 18 days prior to randomization: Days 1, 2, 3 and 16, 17, 18: 150 milligrams (mg) DEM will be taken orally every 6 hours; Days 4 to15: DEM will not be administered.
  Tetracycline (TET): Beginning 22 days prior to the biopsy procedure: Days 1, 2, 3 and 16, 17, 18: 250 mg TET will be taken orally every 6 hours; Days 4 through 15: TET will not be administered.
  Calcium: Approximately 1000 milligrams per day (mg/day) administered orally.
  Vitamin D: Approximately 800 to 1200 International Units per day (IU/day) administered orally.
  Interventions: Drug: Teriparatide; Drug: Demeclocycline; Drug: Tetracycline; Drug: Calcium Supplement; Drug: Vitamin D
- Denosumab (Active Comparator): 60 mg denosumab administered SC once in 6 months.
  DEM: Beginning 18 days prior to randomization: Days 1, 2, 3 and 16, 17, 18: 150 mg DEM will be taken orally every 6 hours; Days 4 to 15: DEM will not be administered.
  TET: Beginning 22 days prior to the biopsy procedure: Days 1, 2, 3 and 16, 17, 18: 250 mg TET will be taken orally every 6 hours; Days 4 through 15: TET will not be administered.
  Calcium: Approximately 1000 mg/day administered orally.
  Vitamin D: Approximately 800 to 1200 IU/day administered orally.
  Interventions: Drug: Denosumab; Drug: Demeclocycline; Drug: Tetracycline; Drug: Calcium Supplement; Drug: Vitamin D

INTERVENTIONS:
Drug: Teriparatide — Administered SC
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: Denosumab — Administered SC
  Arms: Denosumab
Drug: Demeclocycline — Administered orally
Drug: Tetracycline — Administered orally
Drug: Calcium Supplement — Administered orally
Drug: Vitamin D — Administered orally

SUMMARY:
The purpose of this study is to determine how teriparatide or denosumab affects the bone of postmenopausal women with osteoporosis after 3 months of treatment, as determined by a bone biopsy sample taken from the iliac crest (upper part of the pelvis).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women (no vaginal bleeding for at least 2 years prior to screening) with osteoporosis
* Bone mineral density (BMD) T-score of at least -2.5 at femoral neck (FN), total hip (TH), or lumbar spine (LS) (Lumbar vertebrae L1-L4, with at least 2 evaluable vertebrae), with or without atraumatic fracture after menopause, OR
* BMD T-score of at least -1.5 at FN, TH, or LS (L1-L4, with at least 2 evaluable vertebrae), and 1 or more atraumatic fractures after menopause (vertebral or nonvertebral). Nonvertebral fracture sites allowed are wrist, hip, pelvis, rib, humerus, clavicle, leg (femur, tibia, and fibula, excluding ankle)
* Laboratory values for serum calcium, parathyroid hormone (PTH), and alkaline phosphatase must be within the normal reference range

Exclusion Criteria:

* Has an increased risk of osteosarcoma (bone tumor); this includes Paget's disease of bone, a previous bone tumor, or radiation involving the skeleton
* Has an allergy or intolerance to teriparatide or denosumab and/or is a poor candidate for teriparatide or denosumab treatment (investigator should refer to local product prescribing information)
* Has a history of exposure to DEM or TET therapy in the 12 months prior to screening or a known allergy to DEM or TET
* Has a condition that could put the participant at additional risk of an adverse event (AE) due to the bone biopsy procedure (for example, bleeding disorder)
* Has undergone 2 previous iliac crest bone biopsies (1 in each iliac crest)
* Has a 25-hydroxyvitamin D concentration of <10 nanograms per milliliter (ng/mL)
* Has currently active or suspected (within 1 year prior to enrollment) diseases that affect bone metabolism, other than osteoporosis (such as renal osteodystrophy, hyperthyroidism, osteomalacia, or hyperparathyroidism)
* Has a history of certain cancers within 5 years prior to trial entry
* Current or recent (within 1 year prior to enrollment) celiac disease, inflammatory bowel disease, gastric bypass, or other malabsorption syndrome
* Has significantly impaired hepatic or renal function
* Has had treatment with systemic glucocorticoids in doses ≥5 mg/day prednisone/day or equivalent in the 6 calendar months prior to screening
* Has taken any intravenous osteoporosis medication
* Has had prior treatment with other bisphosphonates and not been off of them for a specific period of time before trial entry
* Has participated in any other clinical trial studying teriparatide, PTH, PTH analog, or denosumab, or prior or current treatment with teriparatide, PTH, PTH analog, or denosumab

Ages: 55 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec

REFERENCES:
- [Derived] Dempster DW, Zhou H, Recker RR, Brown JP, Recknor CP, Lewiecki EM, Miller PD, Rao SD, Kendler DL, Lindsay R, Krege JH, Alam J, Taylor KA, Melby TE, Ruff VA. Remodeling- and Modeling-Based Bone Formation With Teriparatide Versus Denosumab: A Longitudinal Analysis From Baseline to 3 Months in the AVA Study. J Bone Miner Res. 2018 Feb;33(2):298-306. doi: 10.1002/jbmr.3309. Epub 2017 Nov 15. PMID 29024120

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Tetracycline (TET) and demeclocycline (DEM) temporarily bind to new bone and are detected as different colors under ultraviolet light in bone biopsy samples. In this study, participants were administered DEM prior to randomization (baseline) and again with TET 22 days prior to bone biopsy obtained 3 months post first dose of study drug.
Groups:
- Teriparatide: Teriparatide: 20-microgram (µg) subcutaneous (SC) injection once daily for 6 months.
  DEM: 150-milligram (mg) tablets administered orally, on the following days, 18 days prior to randomization:
  * Days 1, 2, 3, 16, 17, and 18: 150 mg DEM every 6 hours.
  * Days 4 through 15: DEM was not administered.
  TET: 250-mg capsules administered orally on the following days, 22 days prior to biopsy procedure:
  * Days 1, 2, 3, 16, 17, and 18: 250 mg TET every 6 hours.
  * Days 4 through 15: TET was not administered.
  Calcium Supplements: Approximately 1000 milligrams per day (mg/day) administered orally for 6 months.
  Vitamin D Supplements: Approximately 800 to 1200 International Units per day (IU/day) administered orally for 6 months.
- Denosumab: Denosumab: A single 60-mg SC injection.
  DEM: 150-mg tablets administered orally on the following days, 18 days prior to randomization:
  * Days 1, 2, 3, 16, 17, and 18: 150 mg DEM every 6 hours.
  * Days 4 through 15: DEM was not administered.
  TET: 250-mg capsules administered orally on the following days, 22 days prior to biopsy procedure:
  * Days 1, 2, 3, 16, 17, and 18: 250 mg TET every 6 hours.
  * Days 4 through 15: TET was not administered.
  Calcium Supplements: Approximately 1000 mg/day administered orally for 6 months.
  Vitamin D Supplements: Approximately 800 to 1200 IU/day administered orally for 6 months.
Period: Overall Study
Arm/Group | Teriparatide | Denosumab
Started | 33 | 36
Received at Least 1 Dose of Study Drug | 33 | 36
Completed 3-Month Bone Biopsy | 31 | 35
Completed | 30 | 34
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Sponsor Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug (teriparatide or denosumab).
Groups:
- Teriparatide: Teriparatide: 20-µg SC injection once daily for 6 months.
  DEM: 150-mg tablets administered orally, on the following days, 18 days prior to randomization:
  * Days 1, 2, 3, 16, 17, and 18: 150 mg DEM every 6 hours.
  * Days 4 through 15: DEM was not administered.
  TET: 250-mg capsules administered orally on the following days, 22 days prior to biopsy procedure:
  * Days 1, 2, 3, 16, 17, and 18: 250 mg TET every 6 hours.
  * Days 4 through 15: TET was not administered.
  Calcium Supplements: Approximately 1000 mg/day administered orally for 6 months.
  Vitamin D Supplements: Approximately 800 to 1200 IU/day administered orally for 6 months.
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Denosumab | Total
Number analyzed (Participants) | 33 | 36 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.58 (5.84) | 65.17 (8.32) | 63.45 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 31 | 32 | 63
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 31 | 31 | 62
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 27 | 48
  Canada | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 3 Months in Mineralizing Surface (MS) /Bone Surface (BS) in the Cancellous Compartment (CC) of the Iliac Crest Bone Biopsies
Description: MS /BS is a measure of the proportion of BS on which new mineralized bone is deposited at the time of DEM or TET labeling, and calculated as the sum of the total extent of double label (DL) plus half the extent of single label (SL) divided by BS. At baseline (18 days prior to randomization / study drug administration), DEM was administered (3 days on, 12 days off, 3 days on). 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered (same dosing schedule as DEM). Both DEM and TET temporarily bind to new bone and fluoresce under UV light. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation and a SL or no label (NL) suggested varying degrees of suppression of bone formation.
Time Frame: Baseline, 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with MS/BS measurements in the CC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of BS
Groups:
- Teriparatide: Teriparatide: 20-mcg SC injection once daily for 6 months.
  DEM: 150-mg tablets administered orally, on the following days, 18 days prior to randomization:
  * Days 1, 2, 3, 16, 17, and 18: 150 mg DEM every 6 hours.
  * Days 4 through 15: DEM was not administered.
  TET: 250-mg capsules administered orally on the following days, 22 days prior to biopsy procedure:
  * Days 1, 2, 3, 16, 17, and 18: 250 mg TET every 6 hours.
  * Days 4 through 15: TET was not administered.
  Calcium Supplements: Approximately 1000 mg/day administered orally for 6 months.
  Vitamin D Supplements: Approximately 800 to 1200 IU/day administered orally for 6 months.
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of BS | 12.43 [7.81 to 18.97] | -2.51 [-5.08 to -1.22]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) model with treatment group as the main effect and baseline MS/BS as a covariate

2. Secondary Outcome: Number of Samples With Single or Double Tetracycline Labels, SL and DL, or No Tetracycline Labels in the CC, Endocortical Compartment (EC), Intracortical Compartment (IC) and Periosteal Compartment (PC) of the Iliac Crest Bone Biopsies
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with an assessment of the number of samples with specified labels in the various compartments of the iliac crest.
Measure: Number; unit: Samples
Groups:
- Teriparatide: Teriparatide: 20-mcg SC injection once daily for 6 months.
  DEM: 150-mg tablets administered orally, on the following days, prior to randomization:
  * Days 1, 2, 3, 16, 17, and 18: 150 mg DEM every 6 hours.
  * Days 4 through 15: DEM was not administered.
  TET: 250-mg capsules administered orally on the following days, prior to biopsy procedure:
  * Days 1, 2, 3, 16, 17, and 18: 250 mg TET every 6 hours.
  * Days 4 through 15: TET was not administered.
  Calcium Supplements: Approximately 1000 mg/day administered orally for 6 months.
  Vitamin D Supplements: Approximately 800 to 1200 IU/day administered orally for 6 months.
- Denosumab: Denosumab: A single 60-mg SC injection.
  DEM: 150-mg tablets administered orally on the following days, prior to randomization:
  * Days 1, 2, 3, 16, 17, and 18: 150 mg DEM every 6 hours.
  * Days 4 through 15: DEM was not administered.
  TET: 250-mg capsules administered orally on the following days, prior to biopsy procedure:
  * Days 1, 2, 3, 16, 17, and 18: 250 mg TET every 6 hours.
  * Days 4 through 15: TET was not administered.
  Calcium Supplements: Approximately 1000 mg/day administered orally for 6 months.
  Vitamin D Supplements: Approximately 800 to 1200 IU/day administered orally for 6 months.
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
Samples
  DL and SL, in CC (n=31, 35) | 31 | 24
  DL Only, in CC (n=31, 35) | 0 | 0
  SL Only, in CC (n=31, 35) | 0 | 9
  No Label, in CC (n=31, 35) | 0 | 2
  DL and SL, in EC (n=30, 35) | 30 | 25
  DL Only, in EC (n=30, 35) | 0 | 0
  SL Only, in EC (n=30, 35) | 0 | 6
  No Label, in EC (n=30, 35) | 0 | 4
  DL and SL, in IC (n=30, 35) | 30 | 24
  DL Only, in IC (n=30, 35) | 0 | 0
  SL Only, in IC (n=30, 35) | 0 | 10
  No Label, in IC (n=30, 35) | 0 | 1
  DL and SL, in PC (n=30, 35) | 10 | 1
  DL Only, in PC (n=30, 35) | 0 | 0
  SL Only, in PC (n=30, 35) | 19 | 4
  No Label, in PC (n=30, 35) | 1 | 30
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Fisher Exact — DL and SL, in CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.002, Fisher Exact — SL Only, in CC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.494, Fisher Exact — No Label, in CC
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.001, Fisher Exact — DL and SL, in EC
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.027, Fisher Exact — SL Only, in EC
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.118, Fisher Exact — No Label, in EC
Statistical Analysis 7: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Fisher Exact — DL and SL, in IC
Statistical Analysis 8: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.001, Fisher Exact — SL Only, in IC
Statistical Analysis 9: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p > 0.999, Fisher Exact — No Label, in IC
Statistical Analysis 10: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.002, Fisher Exact — DL and SL, in PC
Statistical Analysis 11: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Fisher Exact — SL Only, in PC
Statistical Analysis 12: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Fisher Exact — No Label, in PC

3. Secondary Outcome: Change From Baseline to 3 Months in MS/BS in the Endocortical Compartment (EC), Intracortical Compartment (IC), and Periosteal Compartment (PC) of the Iliac Crest Bone Biopsies
Description: MS /BS is a measure of the proportion of BS on which new mineralized bone is deposited at the time of DEM or TET labeling and is calculated as the sum of the total extent of DL plus half the extent of SL divided by BS. At baseline (18 days prior to randomization / study drug administration), DEM was administered (3 days on, 12 days off, 3 days on). 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered (same dosing schedule as DEM). Both DEM and TET temporarily bind to new bone and fluoresce under UV light. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation and a SL or NL suggested varying degrees of suppression of bone formation.
Time Frame: Baseline, 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with MS/BS measurements in the specified compartments of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of BS
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 30 | 35
percentage of BS
  EC | 26.12 [13.76 to 47.63] | -2.97 [-5.39 to 0.08]
  IC | 9.39 [4.46 to 19.31] | -6.70 [-12.80 to -3.87]
  PC | 2.40 [0.81 to 7.85] | -0.39 [-1.75 to 0.00]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — EC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — IC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — PC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate

4. Secondary Outcome: MS/BS in the CC, EC, IC and PC of the Iliac Crest Bone Biopsies 3 Months Post First Dose of Study Drug
Description: as for outcome 3
Time Frame: 3 months post first dose of study drug
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: percentage of BS
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of BS
  CC (n=31, 35) | 18.73 [11.13 to 26.64] | 0.96 [0.44 to 1.93]
  EC (n=30, 35) | 39.50 [23.92 to 60.39] | 5.42 [2.63 to 10.15]
  IC (n=30, 35) | 21.69 [15.61 to 30.17] | 3.05 [2.03 to 7.38]
  PC (n=30, 35) | 4.69 [1.24 to 8.98] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — EC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — IC
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — PC

5. Secondary Outcome: Percentage of Bone With Remodeling-Based and Modeling-Based Formations in the CC, EC and PC of the Iliac Crest Bone Biopsies
Description: In this study, post-treatment DLs in the CC, EC, and PC were classified as remodeling-based or modeling-based bone formations which was determined by whether the underlying reversal line was scalloped or smooth and by the collagen fiber orientation. Percentage = (remodeling-based formation units or modeling-based formation units/ total bone formation units) * 100.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with the classification of TET DLs as remodeling-based or modeling-based formation in the specified compartments of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of the total formation unit
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 32
percentage of the total formation unit
  Remodeling-Based Bone Formation in CC (n=31, 32) | 89.02 [86.52 to 92.86] | 90.83 [70.71 to 100.00]
  Modeling-Based Bone Formation in CC (n=31, 32) | 10.98 [7.14 to 13.48] | 9.17 [0.00 to 29.29]
  Remodeling-Based Bone Formation in EC (n=30, 29) | 83.33 [65.00 to 90.00] | 100.00 [80.00 to 100.00]
  Modeling-Based Bone Formation in EC (n=30, 29) | 16.67 [10.00 to 35.00] | 0.00 [0.00 to 20.00]
  Remodeling-Based Bone Formation in PC (n=29, 5) | 0.00 [0.00 to 11.11] | 0.00 [0.00 to 0.00]
  Modeling-Based Bone Formation in PC (n=29, 5) | 100.0 [88.89 to 100.00] | 100.00 [100.00 to 100.00]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.740, Wilcoxon (Mann-Whitney) — Remodeling-Based Bone Formation in the CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.740, Wilcoxon (Mann-Whitney) — Modeling-Based Bone Formation in the CC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — Remodeling-Based Bone Formation in the EC
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — Modeling-Based Bone Formation in the EC
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.661, Wilcoxon (Mann-Whitney) — Remodeling-Based Bone Formation in the PC
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.661, Wilcoxon (Mann-Whitney) — Modeling-Based Bone Formation in the PC

6. Secondary Outcome: Percentage of Mineralizing Surface With Remodeling-Based Formation and Modeling-Based Formation in the CC, EC and PC of the Iliac Crest Bone Biopsies
Description: The percentage of mineralizing surface where post-treatment DLs in the CC, EC, and PC were classified as remodeling-based or modeling based bone formation based on collagen fiber orientation and whether the underlying reversal line was scalloped or smooth.
  Percentage = percentage remodeling- or modeling-based formation units * MS/BS
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with the classification of TET DLs as remodeling- or modeling-based formation in the specified compartments of the iliac crest.
Measure: Median (Full Range); unit: percentage of the total formation unit
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of the total formation unit
  Remodeling-Based Bone Formation in CC (n=31, 35) | 16.67 [0 to 100] | 0.87 [0 to 100]
  Modeling-Based Bone Formation in CC (n=31, 35) | 2.06 [0 to 100] | 0.09 [0 to 100]
  Remodeling-Based Bone Formation in EC (n=30, 35) | 32.92 [0 to 100] | 5.42 [0 to 100]
  Modeling-Based Bone Formation in EC (n=30, 35) | 6.58 [0 to 100] | 0.00 [0 to 100]
  Remodeling-Based Bone Formation in PC (n=30, 35) | 0.00 [0 to 100] | 0.00 [0 to 100]
  Modeling-Based Bone Formation in PC (n=30, 35) | 4.69 [0 to 100] | 0.00 [0 to 100]

7. Secondary Outcome: Percentage of Overfilled Remodeling Sites in the CC, EC and PC of the Iliac Crest Bone Biopsies
Description: The percentage of overfilled remodeling sites in the CC, EC, and PC were defined as the percentage of observed remodeling units in which the second DL (TET) extended beyond the limits of the scalloped reversal line and into the adjacent, previously unresorbed surface of the bone. Percentage = (overfilled remodeling bone formation unit / total bone formation unit) * 100.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy evaluated for overfilled remodeling sites in the specified compartments of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of overfilled remodeling site
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 32
percentage of overfilled remodeling site
  CC (n=31, 32) | 17.74 [10.94 to 23.85] | 0.00 [0.00 to 14.29]
  EC (n=30, 29) | 21.98 [11.11 to 33.33] | 0.00 [0.00 to 14.29]
  PC (n=29, 5) | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — EC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.740, Wilcoxon (Mann-Whitney) — PC

8. Secondary Outcome: Change From Baseline to 3 Months in Label Length Within Each Basic Multicellular Unit (BMU) in the CC, EC, IC and PC of the Iliac Crest Bone Biopsies
Description: BMUs are local groups of osteoblasts and osteoclasts that act in concert to complete a single remodeling cycle. The label length is a measure of the extent of the mineralization front within each BMU in the CC, EC, IC and PC. At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation, and a SL or NL suggested suppression of bone formation.
Time Frame: Baseline, 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with label lengths measured in the specified compartments of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: millimeters (mm)
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 30 | 25
millimeters (mm)
  CC (n=30, 24) | 0.19 [0.13 to 0.22] | 0.05 [0.00 to 0.12]
  EC (n=28, 25) | 0.25 [0.08 to 0.31] | 0.03 [-0.04 to 0.18]
  IC (n=30, 24) | 0.18 [0.16 to 0.25] | 0.02 [-0.07 to 0.11]
  PC (n=4, 1) | 0.12 [-0.02 to 0.60] | 0.10 [0.10 to 0.10]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.004, ANCOVA — EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.850, ANCOVA — PC; ANCOVA model with treatment group as the main effect and baseline as a covariate

9. Secondary Outcome: Change From Baseline to 3 Months in Mineral Apposition Rate (MAR) in the CC, EC, IC and PC of the Iliac Crest Bone Biopsies
Description: MAR is a measure of the linear rate of production of mineralized bone matrix by osteoblasts and is measured by the mean distance between 2 consecutive labels divided by the time interval. At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation, and a SL or NL suggested suppression of bone formation. SL cases were imputed to a value of 0.3 micrometers per day (µm/day) or counted as missing. NL cases were reported as missing.
Time Frame: Baseline, 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with an evaluation of MAR in the CC, EC, IC and PC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: mcm/day
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 34
mcm/day
  DL Only, in CC (n=30, 24) | 0.00 [-0.02 to 0.04] | -0.04 [-0.11 to 0.01]
  DL and Imputed SL, in CC (n=31, 33) | 0.01 [-0.02 to 0.06] | -0.06 [-0.15 to -0.00]
  DL Only, in EC (n=28, 25) | 0.03 [-0.03 to 0.08] | -0.07 [-0.12 to 0.01]
  DL and Imputed SL, in EC (n=29, 31) | 0.03 [-0.03 to 0.08] | -0.09 [-0.16 to 0.00]
  DL Only, in IC (n=30, 24) | 0.20 [0.09 to 0.34] | -0.18 [-0.28 to -0.10]
  DL and Imputed SL, in IC (n=30, 34) | 0.20 [0.09 to 0.34] | -0.22 [-0.33 to -0.12]
  DL Only, in PC (n=4, 1) | 0.05 [-0.14 to 0.11] | -0.04 [-0.04 to -0.04]
  DL and Imputed SL, in PC (n=19, 4) | 0.00 [-0.03 to 0.08] | -0.04 [-0.07 to -0.02]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.004, ANCOVA — DL Only, in CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in the CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL Only, in EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL Only, in IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 7: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.931, ANCOVA — DL Only, in PC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 8: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.549, ANCOVA — DL and Imputed SL, in PC; ANCOVA model with treatment group as the main effect and baseline as a covariate

10. Secondary Outcome: Change From Baseline to 3 Months in Bone Formation Rate/Bone Surface (BFR/BS ) in the CC, EC, IC and PC of the Iliac Crest Bone Biopsies
Description: BFR/BS is the volume of mineralized bone formed per unit surface of bone per unit of time [mm cubed per mm squared per year (mm³/mm²/year)]. At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicates active bone formation, a SL or NL suggests suppression of bone formation. BFR = MAR * (MS/BS). SL cases were imputed to a value of 0.3 mcm/day or counted as missing. NL cases were assigned a value of zero.
Time Frame: Baseline, 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with BFR/BS assessments in the specified compartments of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: mm³/mm²/year
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
mm³/mm²/year
  DL Only, in CC (n=30, 26) | 0.0280 [0.0173 to 0.0426] | -0.0056 [-0.0093 to -0.0021]
  DL and Imputed SL, in CC (n=31, 35) | 0.0275 [0.0143 to 0.0426] | -0.0055 [-0.0094 to -0.0021]
  DL Only, in EC (n=29, 28) | 0.0509 [0.0300 to 0.1105] | -0.0069 [-0.0118 to 0.0002]
  DL and Imputed SL, in EC (n=30, 35) | 0.0501 [0.0300 to 0.1105] | -0.0069 [-0.0123 to -0.0016]
  DL Only, in IC (n=30, 25) | 0.0455 [0.0208 to 0.0654] | -0.0184 [-0.0290 to -0.0103]
  DL and Imputed SL, in IC (n=30, 35) | 0.0455 [0.0208 to 0.0654] | -0.0184 [-0.0290 to -0.0103]
  DL Only, in PC (n=6, 16) | 0.0231 [0.0058 to 0.0369] | 0.0000 [-0.0019 to 0.0000]
  DL and Imputed SL, in PC (n=30, 35) | 0.0015 [0.0008 to 0.0101] | -0.0005 [-0.0019 to 0.0000]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL Only, in CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL Only, in EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL Only, in IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 7: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL Only, in PC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 8: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — DL and Imputed SL, in PC; ANCOVA model with treatment group as the main effect and baseline as a covariate

11. Secondary Outcome: Percentage of Single or Double Tetracycline Labels Per Bone Surface (sLS/BS or dLS/BS) in the CC, EC, IC and PC of the Iliac Crest Bone Biopsies
Description: At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation and a SL or NL suggested suppression of bone formation. Percentage = (Single or double TET labels / BS) *100.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with label surface measured in the specified compartments of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of TET label
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of TET label
  sLS/BS, in CC (n=31, 35) | 15.44 [10.16 to 18.53] | 1.28 [0.66 to 2.62]
  dLS/BS, in CC (n=31, 35) | 10.44 [6.00 to 15.41] | 0.22 [0.00 to 0.79]
  sLS/BS, in EC (n=30, 35) | 24.24 [14.65 to 30.32] | 7.18 [4.13 to 10.58]
  dLS/BS, in EC (n=30, 35) | 28.84 [12.83 to 43.96] | 1.68 [0.00 to 5.08]
  sLS/BS, in IC (n=30, 35) | 15.28 [11.17 to 17.26] | 4.66 [2.54 to 9.57]
  dLS/BS, in IC (n=30, 35) | 14.96 [10.55 to 19.69] | 0.83 [0.00 to 1.87]
  sLS/BS, in PC (n=30, 35) | 9.37 [2.47 to 13.92] | 0.00 [0.00 to 0.00]
  dLS/BS, in PC (n=30, 35) | 0.00 [0.00 to 0.62] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — sLS/BS, in CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — dLS/BS, in CC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — sLS/BS, in EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — dLS/BS, in EC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — sLS/BS, in IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — dLS/BS, in IC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 7: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — sLS/BS, in PC; ANCOVA model with treatment group as the main effect and baseline as a covariate
Statistical Analysis 8: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.028, ANCOVA — dLS/BS, in PC; ANCOVA model with treatment group as the main effect and baseline as a covariate

12. Secondary Outcome: Percentage Change From Baseline to 1, 3, and 6 Months in Intact Parathyroid Hormone (PTH)
Description: PTH regulates calcium and phosphate metabolism in bone and kidney, and is typically measured in serum using the intact PTH assay. Percentage = (PTH value at specified time points - PTH value at baseline) / PTH value at baseline * 100.
Time Frame: Baseline, 1, 3, and 6 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had serum PTH assessed at baseline and the specified time points.
Measure: Median (Inter-Quartile Range); unit: percentage change in PTH
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 28 | 34
percentage change in PTH
  1 month (n=28, 34) | -26.89 [-52.28 to -12.81] | 72.24 [29.87 to 119.53]
  3 months (n=18, 28) | -32.16 [-38.80 to -10.17] | 46.68 [0.21 to 78.87]
  6 months (n=27, 33) | -40.18 [-63.29 to -10.14] | 30.40 [0.00 to 60.57]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 6 months

13. Secondary Outcome: Percentage Change From Baseline to 1, 3, and 6 Months in Serum Procollagen Type I N-terminal Propeptide (P1NP)
Description: P1NP is a marker of bone turnover and is a measure of bone formation. Percentage = (P1NP value at specified time points - P1NP value at baseline) / P1NP value at baseline * 100.
Time Frame: Baseline, 1, 3, and 6 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had serum P1NP measurements at baseline and the specified time points.
Measure: Median (Inter-Quartile Range); unit: percentage change in P1NP
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 33 | 34
percentage change in P1NP
  1 month (n=33, 34) | 134.38 [93.77 to 194.96] | -11.56 [-26.87 to -0.73]
  3 months (n=22, 29) | 213.15 [104.94 to 325.78] | -66.64 [-73.46 to -59.26]
  6 months (n=31, 32) | 284.22 [180.86 to 536.92] | -68.24 [-75.31 to -55.31]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 6 months

14. Secondary Outcome: Percentage Change From Baseline to 1, 3, and 6 Months in Serum Osteocalcin
Description: Osteocalcin is a marker of bone turnover and a measure of osteoblast function. Percentage = (osteocalcin value at specified time points - osteocalcin value at baseline) / (osteocalcin value at baseline) * 100.
Time Frame: Baseline, 1, 3, and 6 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had serum osteocalcin measured at baseline and the specified time points.
Measure: Median (Inter-Quartile Range); unit: percentage change in osteocalcin
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 33
percentage change in osteocalcin
  1 month (n=31, 33) | 90.53 [61.19 to 127.56] | -6.56 [-16.83 to 7.34]
  3 months (n=20, 29) | 123.66 [83.20 to 174.59] | -45.70 [-52.20 to -38.60]
  6 months (n=29, 31) | 187.29 [131.24 to 290.30] | -50.53 [-59.89 to -37.15]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 6 months

15. Secondary Outcome: Percentage Change From Baseline to 1, 3, and 6 Months in Serum Carboxyterminal Cross-Linking Telopeptide of Type I Collagen (CTX)
Description: CTX is a marker of bone turnover and is a measure of bone resorption. Percentage = (CTX value at specified time points - CTX value at baseline) / (CTX value at baseline) * 100.
Time Frame: Baseline, 1, 3, and 6 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and serum CTX measured at baseline and the specified time points.
Measure: Median (Inter-Quartile Range); unit: percentage change in CTX
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 33
percentage change in CTX
  1 month (n=31, 33) | 6.09 [-21.35 to 43.75] | -90.70 [-92.11 to -87.50]
  3 months (n=21, 29) | 73.04 [33.33 to 140.00] | -90.77 [-92.59 to -85.92]
  6 months (n=29, 33) | 89.13 [50.00 to 220.29] | -82.50 [-86.96 to -60.00]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — 6 months

16. Secondary Outcome: Activation Frequency (Ac.f) in the CC, EC and IC of the Iliac Crest
Description: Ac.f is the probability of new remodeling cycles initiated on the BS per year. Ac.f = (BFR/BS) / wall thickness. At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation and a SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing. NL cases were assigned a value of zero.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with Ac.f assessments in the CC, EC and IC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: new cycles per year
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
new cycles per year
  DL Only, in CC (n=31, 26) | 1.41 [0.88 to 2.02] | 0.10 [0.04 to 0.20]
  DL and Imputed SL, in CC (n=31, 35) | 1.41 [0.88 to 2.02] | 0.06 [0.02 to 0.14]
  DL Only, in EC (n=30, 29) | 2.77 [1.48 to 4.31] | 0.35 [0.19 to 0.62]
  DL and Imputed SL, in EC (n=30, 35) | 2.77 [1.48 to 4.31] | 0.34 [0.09 to 0.59]
  DL Only, in IC (n=30, 25) | 1.88 [1.13 to 2.48] | 0.17 [0.11 to 0.36]
  DL and Imputed SL, in IC (n=30, 35) | 1.88 [1.13 to 2.48] | 0.12 [0.06 to 0.27]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL Only, in CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL and Imputed SL, in CC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL Only, in EC
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL and Imputed SL, in EC
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL Only, in IC
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL and Imputed SL, in IC

17. Secondary Outcome: Adjusted Apposition Rate (Aj.AR) in the CC, EC and IC of the Iliac Crest
Description: Aj.AR is MAR averaged over the entire osteoid surface and in a steady state is an estimate of the mean rate of matrix apposition. At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation and a SL or NL suggested suppression of bone formation. BFR = MAR * (MS/BS). SL cases were imputed to a value of 0.3 µm/day or counted as missing. NL cases were counted as missing.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with Aj.AR assessments in the CC, EC and IC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: µm/day
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 33
µm/day
  DL Only, in CC (n=31, 24) | 0.58 [0.46 to 0.67] | 0.21 [0.09 to 0.48]
  DL and Imputed SL, in CC (n=31, 33) | 0.58 [0.46 to 0.67] | 0.14 [0.08 to 0.33]
  DL Only, in EC (n=30, 25) | 0.76 [0.56 to 0.88] | 0.65 [0.41 to 0.82]
  DL and Imputed SL, in EC (n=30, 30) | 0.76 [0.56 to 0.88] | 0.58 [0.22 to 0.81]
  DL Only, in IC (n=30, 24) | 1.03 [0.88 to 1.18] | 0.58 [0.26 to 0.83]
  DL and Imputed SL, in IC (n=30, 33) | 1.03 [0.88 to 1.18] | 0.35 [0.19 to 0.73]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — DL Only, in CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL and Imputed SL, in CC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.214, Wilcoxon (Mann-Whitney) — DL Only, in EC
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney) — DL and Imputed SL, in EC
Statistical Analysis 5: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL Only, in IC
Statistical Analysis 6: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — DL and Imputed SL, in IC

18. Secondary Outcome: Percentage of Osteoid Volume (OV)/Bone Volume (BV) in the CC of the Iliac Crest
Description: OV is the percentage of a given volume of bone tissue that consists of new unmineralized bone matrix (osteoid). Percentage = (OV/BV) *100.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with an assessment of OV/BV in the CC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of BV
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of BV | 2.58 [1.67 to 3.51] | 0.39 [0.17 to 0.65]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Percentage of Osteoid Surface (OS)/Bone Surface (BS) in the CC, EC and IC of the Iliac Crest
Description: OS is the percentage of the entire trabecular BS that is covered by osteoid. Percentage = (OS / BS) *100.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with the assessment of OS/BS in the CC, EC and IC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of BS
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of BS
  CC (n=31, 35) | 20.51 [12.50 to 24.13] | 3.46 [2.05 to 5.40]
  EC (n=30, 35) | 30.85 [21.47 to 48.02] | 6.95 [2.82 to 10.88]
  IC (n=30, 35) | 17.81 [11.89 to 22.50] | 4.34 [2.07 to 6.17]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — EC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — IC

20. Secondary Outcome: Osteoid Thickness (O.Th) in the CC, EC and IC of the Iliac Crest
Description: O.Th is a measure of the average thickness of osteoid seams.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with an O.Th assessment in the CC, EC and IC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: micrometers (mcm)
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
micrometers (mcm)
  CC (n= 31, 35) | 6.12 [5.52 to 6.71] | 3.78 [3.49 to 4.18]
  EC (n= 30, 35) | 6.99 [5.61 to 7.99] | 4.33 [3.49 to 4.78]
  IC (n= 30, 35) | 7.08 [6.15 to 7.92] | 4.68 [3.68 to 5.13]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — EC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — IC

21. Other Pre Specified Outcome: Average Length of DLs in the CC, EC, IC and PC of the Iliac Crest
Description: The length of TET DLs is a measure of the extent of bone formation in each compartment within individual remodeling units and is measured in mm. At baseline (18 days prior to randomization / study drug administration), DEM was administered. 22 days prior to the biopsy procedure (biopsy obtained 3 months post first dose of study drug), TET was administered. New bone in the biopsy was seen as the amount of bone between the 2 fluorescently DEM- or TET-labeled lines under a microscope. A DL indicated active bone formation.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with an assessment of DL length in the various compartments of the iliac crest.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 25
mm
  DL, in CC (n=31, 24) | 0.40 (0.08) | 0.31 (0.10)
  DL, in EC (n=30, 25) | 0.48 (0.15) | 0.35 (0.20)
  DL, in IC (n=30, 24) | 0.43 (0.11) | 0.27 (0.12)
  DL, in PC (n=10, 1) | 0.38 (0.41) | 0.32 (NA) — n=1
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — Average length of DLs in the CC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.004, ANCOVA — Average length of double labels in EC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, ANCOVA — Average length of double labels in IC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate
Statistical Analysis 4: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.850, ANCOVA — Average length of double labels in the PC; ANCOVA model with treatment group as the main effect and baseline MS/BS as a covariate

22. Secondary Outcome: Wall Thickness (W.Th) in the CC, EC and IC of the Iliac Crest
Description: W.Th is the distance from the cement line to the marrow space of completed trabecular bone packets.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with a W. Th assessment in the CC, EC and IC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
µm
  CC (n=31, 35) | 26.29 [25.58 to 27.84] | 24.03 [22.79 to 25.23]
  EC (n=30, 35) | 31.88 [29.75 to 32.99] | 30.08 [27.61 to 32.03]
  IC (n=30, 35) | 38.25 [33.87 to 39.84] | 37.80 [34.61 to 40.15]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney) — EC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p = 0.678, Wilcoxon (Mann-Whitney) — IC

23. Secondary Outcome: Percentage of Eroded Surface/Bone Surface (ES/BS) in the CC, EC and IC of the Iliac Crest
Description: ES/BS is the fraction of the entire trabecular surface occupied by resorption bays, including both those with and without osteoclasts. It is an indicator of bone resorption. Percentage = (ES/BS) *100.
Time Frame: 3 months post first dose of study drug
Population: Randomized participants who received at least 1 dose of study drug and had an evaluable 3-month bone biopsy with ES/BS assessed in the CC, EC and IC of the iliac crest.
Measure: Median (Inter-Quartile Range); unit: percentage of BS
Arm/Group | Teriparatide | Denosumab
Number analyzed (Participants) | 31 | 35
percentage of BS
  CC (n=31, 35) | 3.73 [2.95 to 6.05] | 1.52 [0.92 to 2.87]
  EC (n=30, 35) | 3.79 [2.79 to 6.25] | 1.65 [0.78 to 2.47]
  IC (n=30, 35) | 11.19 [7.37 to 13.71] | 1.27 [0.90 to 3.82]
Statistical Analysis 1: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — CC
Statistical Analysis 2: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — EC
Statistical Analysis 3: Comparison: Teriparatide vs Denosumab; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — IC

ADVERSE EVENTS:
Arm/Group | Teriparatide | Denosumab
Serious Adverse Events (participants affected / at risk) | 2/33 | 2/36
Other Adverse Events (participants affected / at risk) | 27/33 | 23/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=33) | Denosumab (N=36)
Chest pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=33) | Denosumab (N=36)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 2 (2) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 10 (10) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 2 (2) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Spider vein (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days